CLINICAL TRIAL: NCT04099758
Title: One-session Mindfulness of the Breath Meditation Practice: A Randomized Controlled Study of the Effects on State Hope and State Gratitude
Brief Title: A Study of the Effects of a One-session Mindfulness of the Breath Meditation Practice on State Hope and State Gratitude in the General Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S_Strohmaier_22_07_2019
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomized controlled study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomised and complete the study, including outcome measures, through an automated online programme, without involvement of the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness of the breath meditation (Experimental): 10 minute mindfulness of the breath meditation practice delivered online via audio-recording.
  Interventions: Behavioral: Mindfulness of the breath meditation
- Audio-recording control (Placebo Comparator): 10 minute non-fiction audio-recording delivered online
  Interventions: Behavioral: Audio-recording control

INTERVENTIONS:
Behavioral: Mindfulness of the breath meditation — A 10-minute mindfulness of the breath meditation practice
  Arms: Mindfulness of the breath meditation
Behavioral: Audio-recording control — 10 minute non-fiction audio-recording delivered online
  Arms: Audio-recording control

SUMMARY:
This study aims to examine whether a brief mindfulness of the breath meditation practice is more helpful than listening to an audio recording in relation to improving hope and gratitude in the general population.

DETAILED DESCRIPTION:
This one-session online study will randomise members of the general public to either 1) a mindfulness of the breath meditation practice lasting 10 minutes or 2) an audio-recording control of the same length. State measures of mindfulness, hope and gratitude will be taken immediately before (baseline) and after the intervention/control. In addition, the study will also measure trait mindfulness at baseline.The primary hypothesis is that engaging in a brief mindfulness practice will result in beneficial changes in state hope compared to control. Other hypotheses are that: engaging in a brief mindfulness practice will result in beneficial changes in state gratitude compared to control; that the effect of mindfulness practice on state hope will be statistically mediated by change in state mindfulness; that the effect of mindfulness practice on state gratitude will be statistically mediated by change in state mindfulness; and that baseline trait mindfulness will statistically moderate the effect of mindfulness practice on change in state mindfulness in the above mentioned mediation models (i.e. that moderated mediation will be observed).

ELIGIBILITY:
Inclusion Criteria:

* Members of the general public.
* Adequate understanding of spoken and written English.
* Internet access.

Exclusion Criteria:

-Currently experiencing very severe problems with their mental health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post-intervention on the State Hope Scale (SHS). | Baseline (0 minutes), post-intervention (10 minutes).
  The SHS is a 6-item self-report measure of state hope. The total score on SHS ranges from 8 to 48 , with higher score indicating greater state hope.

SECONDARY OUTCOMES:
Change from baseline to post-intervention on the Gratitude Adjective Checklist (GAC). | Baseline (0 minutes), post-intervention (10 minutes).
  The GAC is a 3-item self-report measure of state gratitude. The total score on GAC ranges from 3 to 15, with higher score indicating greater state gratitude.

OTHER OUTCOMES:
Change from baseline to post-intervention on the Toronto Mindfulness Scale (TMS). | Baseline (0 minutes), post-intervention (10 minutes).
  The TMS is a 13-item self-report measure of state mindfulness that produces scores for curiosity and decentering. The curiosity score ranges from 0 to 24, the decentering score from 0 to 28, and the total score from 0 to 52, with higher scores indicating greater curiosity, decentering and overall state mindfulness respectively.
Five Factor Mindfulness Questionnaire -15 item version (FFMQ-15) | Baseline (0 minutes)
  The FFMQ-15 is a 15-item measure of trait mindfulness. It will be administered at baseline only. The total score on the FFMQ-15 ranges from 15 to 75, with higher score indicating greater trait mindfulness. (Note that the observe subscale will be excluded from the calculation of the total score, as recommended in https://doi.org/10.1002/jclp.21865 and http://dx.doi.org/10.1037/pas0000263 producing a total score between 12 and 60).
Bespoke manipulation check questionnaire. | Post-intervention (10 minutes)
  Participants rate the extent to which they paid attention during the intervention and followed the guidance on 0 - 10 scales, with higher scores indicating greater compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Strohmaier, BA, MSc, Principal Investigator — Canterbury Christ Church University; Fergal Jones, PhD, PsychD, Study Director — Canterbury Christ Church University; James Cane, PhD, Study Director — Canterbury Christ Church University
Locations (1):
- Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom